CLINICAL TRIAL: NCT02054936
Title: Evaluation of Wound Drainage Following Rivaroxaban (Xarelto) or Warfarin (Coumadin) for Post op Venous Thromboembolism (VTE) Prophylaxis, After Knee or Hip Arthroplasty a Randomized Study.
Brief Title: Evaluation of Wound Drainage After Knee or Hip Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in standard of care, no possibility of recruitment
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Andrew Urquhart, M.D. Service Chief Clinical Associate Professor, Orthopaedic Surgery Hip and Knee Replacement, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00062541
Record Dates: First submitted 2014-01-23; First posted 2014-02-04 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Complications; Arthroplasty
MeSH Terms: interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivaroxaban (Xarelto) (Active Comparator): Rivaroxaban dosing will be 10mg once daily beginning on postoperative day 1 for a duration of 30 days.
  Interventions: Drug: Rivaroxaban (Xarelto)
- Warfarin (Coumadin) (Active Comparator): Warfarin dosing will be titrated to achieve an INR of 2-3 and dosing will begin on postoperative day 1 for a duration of 30 days.
  Interventions: Drug: Warfarin (Coumadin)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto) — To date there has been little attention to evaluating differences in wound complications following TJA among patients treated with rivaroxaban compared to warfarin.
  Arms: Rivaroxaban (Xarelto)
Drug: Warfarin (Coumadin) — To date there has been little attention to evaluating differences in wound complications following TJA among patients treated with rivaroxaban compared to warfarin.
  Arms: Warfarin (Coumadin)

SUMMARY:
To compare side effects and complications relating to use of warfarin or rivaroxaban, tolerance and/or toxicity of these two agents such as drop in hemoglobin post operatively, extent of bruising, quantity of wound drainage, duration of drainage, wound swelling, sub and supra-therapeutic prothrombin times, need for transfusion, and patient tolerance in two randomized groups. Return visits to the operating room, length of stay, and VTE rates will also be compared.

ELIGIBILITY:
Inclusion Criteria:

* All patients over the age of 18 undergoing primary hip or knee replacement by Dr. Urquhart or Dr. Hallstrom.

Exclusion Criteria:

* Patients with a contraindication to pharmacologic VTE prophylaxis such as hemophilia, Plavix use, active bleeding or prior reaction to warfarin or rivaroxaban, nursing mothers, hepatic disease, GFR <30, use of more than 200mg of aspirin daily, and inability to continue medication or lab monitoring after hospital discharge known preoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Number of days until a dry wound | 90 days
  Comparative wound oozing time between patients receiving Rivaroxaban and those receiving Warfarin will be measured. Wound will be defined as actively draining if the gauze covering the wound is wet to the edges or if fluid is noted to be originating from the surgical site. The nursing staff will record the wound drainage during the hospital stay and the patient will be instructed in self assessment upon discharge using the patient diary.Wound drainage will be recorded twice daily. Time when the wound appeared dry will be noted.
Amount and character of wound drainage | 90 days
  Wound assessments, including photographs, will occur by a research team member blinided to the anticoagulant being used at three set points; 2 days, 2 weeks, and 6 weeks postoperatively.

SECONDARY OUTCOMES:
Number of days in the hospital postoperatively. | 90 days
  How many days patient is in hospital postoperatively will be noted
Incidence of wound infection | 90 days
  Presence or absence of clinical infection will be noted according to ASEPSIS criteria.
Incidence of additional operations | 90 days
  Additional operations include irrigation and debridement and or revision

OTHER OUTCOMES:
Survey assessments | 90 days
  Satisfaction and activity combined scores from the UCLA Activity Score and the PROMIS Survey at 90 days will be compared to UCLA Activity Score and PROMIS Survey at preoperative visit

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Urquhart, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States